CLINICAL TRIAL: NCT04875000
Title: Effect of Arginine and Nano-hydroxyapatite Solutions on Hypersensitivity and Color Changes of Bleached Enamel: a Randomized Controlled Trial
Brief Title: Hypersensitivity and Color Changes of Bleached Teeth Using Different Remineralizing Agents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2433042021
Record Dates: First submitted 2021-04-24; First posted 2021-05-06 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-04

CONDITIONS: Tooth Hypersensitivity
Keywords: Teeth bleaching; Remineralizing agents; Arginine solution; Nano-hydroxyapatite solution; Hypersensitivity; Color changes
MeSH Terms: conditions — Dentin Sensitivity; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Parallel interventional study model
Who Masked: Participant
Masking Description: None of the participants is aware of the remineralizing agent to be applied to his/her teeth after bleaching
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- UltraEZ (Active Comparator): Group of patients randomly assigned to receive the the application of the commercial fluoride remineralizing and desensitizing agent "UltraEZ (Ultradent Products, Inc, South Jordan, UT, USA)" after teeth bleaching
  Interventions: Other: Remineralizing agent I application
- Arginine (Experimental): Group of patients randomly assigned to receive the the application of the 2.5% arginine solution after teeth bleaching
  Interventions: Other: Remineralizing agent II application
- Nano-hydroxyapatite (Experimental): Group of patients randomly assigned to receive the application of the 2.5% nano-hydroxyapatite solution after teeth bleaching
  Interventions: Other: Remineralizing agent III application

INTERVENTIONS:
Other: Remineralizing agent I application — Application of UltraEZ remineralizing agent to the bleached teeth
  Arms: UltraEZ
Other: Remineralizing agent II application — Application of 2.5% arginine solution to the bleached teeth
  Arms: Arginine
Other: Remineralizing agent III application — Application of 2.5% nano-hydroxyapatite solution to the bleached teeth
  Arms: Nano-hydroxyapatite

SUMMARY:
The aim of this in vivo study is to evaluate the post-bleaching enamel hypersensitivity and the possible color changes following the application of arginine and nano-hydroxyapatite remineralizing solutions after enamel bleaching using an in-office chemical bleaching agent. A commercial Fluoride remineralizing and desensitizing agent will be used as the control group. Following bleaching of the anterior teeth and then the application of the different tested remineralizing agents; the patients will be assessed for post-bleaching hypersensitivity using the visual analogue scale (VAS) to describe the severity of the hypersensitivity from mild to moderate to severe. On the other hand, the baseline shade and post-bleaching color changes will be evaluated using a shade guide. The data will be collected and tabulated then the statistical analysis will be performed.

The null hypothesis is that the different tested remineralizing agents will have a similar effect on the post-bleaching teeth hypersensitivity & the color changes of the bleached teeth.

DETAILED DESCRIPTION:
Recently, there has been several patients that favor the in-office bleaching technique due to its quick and satisfying aesthetic outcome, nevertheless clinical research reported some clinical adverse effects. Teeth hypersensitivity is the most common adverse effect of teeth bleaching. It was suggested that hydrogen peroxide can pass to the pulp through enamel and dentin to create an inflammatory reaction or directly stimulate the neural receptors triggering pain sensation.

It was reported that tooth sensitivity during bleaching has a range of 18-78%. Usually, teeth hypersensitivity subsides upon accomplishment of the bleaching procedure, but occasionally it may cause the patient to withdraw from form the treatment session. Different methods and approaches with a varying rate of success have been advocated to reduce teeth sensitivity, such as decreasing the rate of application, using different desensitizing agents before or after bleaching procedure, desensitizing agent incorporation into the bleaching gel, and decreasing the concentration of bleaching agent. In this context, the efficacy of desensitizing obliteration agents to prevent and treat the post-bleaching hypersensitivity has been investigated in many clinical trials presenting promising results. These obliterating agents can enhance the enamel mineral content, impeding hydrogen peroxide infiltration to the nerve endings and thereby hypersensitivity is much reduced or even eliminated.

Study design:

This randomized clinical study will use the "excel sheet" for randomization and assigning the subjects into the respective test groups.

All the included subjects will sign an informed consent before participating in this clinical study, in full accordance with the World Medical Association Declaration of Helsinki.

Settings and locations:

From the pre-determined inclusion and exclusion criteria, a total of 33 volunteers will be enrolled for the study. The clinical study will be performed from March 2021, through June 2021, in the outpatient dental clinic at the National Research Centre in Egypt.

Sample size calculation:

An equivalence test of means using two one-sided tests based on data from a previous study resulted in a design of 11 patient in each group (control and treatment groups) as minimum sample sizes and will achieves 92% power at a 5.0% significance level when the true difference between the Visual Analogue Scale (VAS) means is 0.3, the standard deviation is 0.3, and the equivalence limits are -0.7 and 0.7.

Tested materials:

The materials to be used in the study will be: an in-office hydrogen peroxide chemical-activated bleaching kit: Opalescence™ Boost™ 40% hydrogen peroxide Tooth Whitening System (Ultradent Products, Inc., South Jordan, UT, USA) and three desensitizing agents: a commercially available UltraEZ desensitizing gel (Ultradent Products, Inc., South Jordan, UT, USA) and 2.5% concentration of arginine and nano-Hydroxy apatite solutions.

Sample grouping:

The enrolled 33 participants will be randomly divided into three groups (n=11) according to the "Coin-Toss method", representing the investigated remineralizing and desensitizing agent to be received after bleaching of their maxillary and mandibular anterior teeth with a 40% hydrogen peroxide in-office chemical-activated bleaching agent as follows:

Group I : UltraEZ desensitizing gel application after bleaching (control). Group II : 2.5% Arginine solution application after bleaching. Group III: 2.5% nano-hydroxyapatite solution application after bleaching.

In-office teeth bleaching:

Pre-operative hypersensitivity will be determined and recorded for all enrolled subjects using the VAS method.

Baseline shade color of the predetermined teeth will be recorded using Classical VITAPAN shade guide.

The in-office bleaching procedure will be performed using Opalescence™ Boost™ 40% Tooth Whitening System (Ultradent Products, Inc., South Jordan, Utah, USA) chemical bleaching agent according to the manufacturer instructions.

Preparation of arginine and nano-hydroxyapatite solutions:

Two and a half g of arginine powder (Sigma-Aldrich, St. Louis, MO, USA), and 2.5 g of nano-hydroxyapatite powder (Sigma-Aldrich, St. Louis, MO, USA) will be weighed with a digital balance then mixed with 100 ml of distilled water to obtain a 2.5%-concentration of arginine and nano-hydroxyapatite solutions.

Application of the remineralizing agents:

A commercially available fluoride agent "UltraEZ gel (Ultradent Products, Inc., South Jordan, UT, USA)" will be applied to the teeth of the assigned patients of Group I and left undisturbed for 20 min as recommended by the manufacturer. Then the patients will be instructed to rinse their teeth thoroughly with water. The 2.5% prepared solutions of arginine and nano-hydroxyapatite will be applied to the bleached teeth of the assigned patients of Group II and Group III respectively, using micro brushes in a generous amount to the labial surfaces of the bleached teeth and left undisturbed for 20 min. Then the patients will be instructed to rinse their teeth thoroughly with water.

Post-operative hypersensitivity evaluation:

The post-operative hypersensitivity of the bleached maxillary anterior teeth will be recorded immediately after bleaching then once again after application of the remineralizing agents at the same session. Tooth sensitivity will be evaluated using a 3-way syringe at 5 to 10 cm distance using the Visual Analogue Scale (VAS). Whereby, readings from 0-10. Zero denoting no sensitivity, 1-3 is presented as mild, 4-7 is presented as moderate and 8-10 is presented as severe sensitivity. After that, it will be recorded on daily bases for the first week by the participants who will be asked to bring their records in the follow-up sessions. Then the postoperative hypersensitivity will be evaluated in-office every week for a 3-week follow-up period using the VAS scoring system. All the readings will be recorded in a self-structured proforma.

Post-operative color evaluation:

The post-bleaching shades of the maxillary anterior teeth will be recorded immediately after bleaching, then once again after application of the desensitizing agents at the same session. Afterwards, it will be recorded every week for a 3-week follow-up period using VITAPAN classical A1-D4® shade guide at the middle third of the anterior maxillary teeth. The 16 tabs of the VITAPAN classical shade guide were arranged in descending numerical order regarding the value from B1 to C4. Then these values were converted into code numbers using a conversion table.

ELIGIBILITY:
Inclusion Criteria:

* Participants of 18-55 years old
* Participants with good general and oral health.
* Participants did not undergo any bleaching procedure before.
* Participants with caries-free maxillary six anterior teeth without any restorations.
* Participants do not suffer of periodontal diseases.
* Participants willing to assess and sign the informed consent form.

Exclusion Criteria:

* Participants with anterior restorations.
* Participants with dental prosthesis of the anterior teeth.
* Participants with orthodontics brackets.
* Participants with severe internal teeth discoloration as in cases of tetracycline stains, fluorosis or non-vital teeth.
* Smoking participants.
* Breastfeeding and pregnant women.
* Participants with gingival and bone recession.
* Participants with dental erosion, dentin exposure, and cracked teeth or any other pathologic condition that may elicit teeth sensitivity.
* Participants having their teeth bleached.
* Participants taking analgesic or anti-inflammatory drugs.
* Participants with bruxism habits are excluded from the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Teeth Hypersensitivity change | Baseline to 3-week follow up period.
  Evaluation of the change in the pre- and post-bleaching teeth hypersensitivity using the Visual Analogue Scale method (VAS) to describe the severity of the hypersensitivity from mild to moderate to severe. Whereby, readings from 0-10. Zero denoting no sensitivity, 1-3 is presented as mild, 4-7 is presented as moderate and 8-10 is presented as severe sensitivity by the description of each one of the participants using a printed chart.

SECONDARY OUTCOMES:
Color change | Baseline to 3-week follow up period.
  Evaluation of the pre- and post-bleaching teeth color change using the VITA classical shade guide at the middle third of the anterior maxillary teeth. The 16 tabs of the VITAPAN classical shade guide will be arranged in descending numerical order regarding the value from B1 to C4. These values will be converted into code numbers using a conversion table.

CONTACTS AND LOCATIONS:
Overall Officials: Lamiaa M Moharam, Ass. Prof, Principal Investigator — National Research Centre, Egypt
Locations (1):
- National Research Centre, Cairo, Giza Governorate, Egypt

REFERENCES:
- [Background] Soares DG, Basso FG, Pontes EC, Garcia Lda F, Hebling J, de Souza Costa CA. Effective tooth-bleaching protocols capable of reducing H(2)O(2) diffusion through enamel and dentine. J Dent. 2014 Mar;42(3):351-8. doi: 10.1016/j.jdent.2013.09.001. Epub 2013 Sep 19. PMID 24056046
- [Background] Browning WD, Chan DC, Myers ML, Brackett WW, Brackett MG, Pashley DH. Comparison of traditional and low sensitivity whiteners. Oper Dent. 2008 Jul-Aug;33(4):379-85. doi: 10.2341/07-134. PMID 18666494
- [Background] Cardoso PC, Reis A, Loguercio A, Vieira LC, Baratieri LN. Clinical effectiveness and tooth sensitivity associated with different bleaching times for a 10 percent carbamide peroxide gel. J Am Dent Assoc. 2010 Oct;141(10):1213-20. doi: 10.14219/jada.archive.2010.0048. PMID 20884923
- [Background] Pintado-Palomino K, Peitl Filho O, Zanotto ED, Tirapelli C. A clinical, randomized, controlled study on the use of desensitizing agents during tooth bleaching. J Dent. 2015 Sep;43(9):1099-1105. doi: 10.1016/j.jdent.2015.07.002. Epub 2015 Jul 6. PMID 26159384
- [Background] Borges BC, Borges JS, de Melo CD, Pinheiro IV, Santos AJ, Braz R, Montes MA. Efficacy of a novel at-home bleaching technique with carbamide peroxides modified by CPP-ACP and its effect on the microhardness of bleached enamel. Oper Dent. 2011 Sep-Oct;36(5):521-8. doi: 10.2341/11-013-L. Epub 2011 Aug 5. PMID 21819199